CLINICAL TRIAL: NCT04205422
Title: Biphasic Intermittent Positive Airway Pressure Versus Airway Pressure Release Ventilation in Critically Ill Trauma Patients: Metabolic Demands and Respiratory Mechanics
Brief Title: Effect of Two Modes of Mechanical Ventilation on Metabolic Demands and Respiratory Mechanics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelbaky Abdelrahman, assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Anesthesia 25
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Mechanical Ventilation
Keywords: metabolic requirements; respiratory mechanics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIPAP group (Active Comparator): Biphasic Intermittent Positive Airway Pressure group
  Interventions: Procedure: BIPAP
- APRV group (Active Comparator): Airway Pressure Release Ventilation group:
  Interventions: Procedure: APRV

INTERVENTIONS:
Procedure: BIPAP — Biphasic Intermittent Positive Airway Pressure
  Arms: BIPAP group
Procedure: APRV — Airway Pressure Release Ventilation
  Arms: APRV group

SUMMARY:
Adequate supply of energy is an essential part of the overall treatment of critically ill patients and adjustment of energy requirements of patients is important clinical evolution .The adequate assessment of energy expenditure is the basis of effective nutri¬tional planning.

DETAILED DESCRIPTION:
Inappropriate energy supply, may cause important complications that affect the progression of the disease, especially in critically ill patients receiving mechanical ventilation. Mechanically ventilated patients make a considerable respiratory muscle effort that is not always decreased by intermittent positive pressure ventilation.

No work of breathing is observed in patients under controlled mechanical ventilation who are receiving drugs for sedation and muscle paralysis. In this situation, the work of breathing is carried out by the ventilator which initiates the ventilation cycle, and patients are spared the inspiratory efforts. Conversely, in assisted ventilation modes, the patient has to make a considerable inspiratory effort before a ventilation cycle initiates, and there is no airflow up to the moment when the effective sensitivity threshold is reached by the ventilator. Therefore, the choice of ventilation mode may determine differences in energy expenditure.

Some studies found that in patients on mechanical ventilation, weight, height, body temperature, type of mechanical ventilation, and type of medication received influenced the REE Acute hypoxemic respiratory failure is a common reason for patients to be admitted to the intensive care unit (ICU). An international study showed an incidence of acute respiratory distress syndrome (ARDS) of 10.4% in ICU critically ill trauma patients with an hospital mortality reaching 46.1% for most severe cases. A protective ventilation strategy using low tidal vol-ume (LTV) and a plateau pressure lower than 30 cmH2O is widely accepted to limit ventilator-induced lung injury, and it currently represents the intervention able to reduce mortality supported by the strongest evidences. Airway pressure release ventilation (APRV) was described for the first time by Stock and Downs and consists in a time-triggered, pressure-limited and time-cycled ventilation mode in which the pressure was alternated from a high level (Phigh) applied for a prolonged time (Thigh) to maintain adequate lung volume and alveo-lar recruitment, to a low level (Plow) for a short period of time (Tlow) where most of ventilation and CO2 removal occurs. In contrast to pressure-controlled inverse-ratio ventilation, APRV uses a release valve that allows spontaneous breathing during any phase of respiratory cycle. The rationale behind this approach is to maintain a pressure above the closing pressure of recruitable alveoli for a sustained time, limiting the release time to allow CO2 removal but avoiding de-recruitment. Another conceptual advantage to APRV over controlled modes is the preservation of spontaneous breathing, which may pro-mote a redistribution of aeration to the dependent lung regions, less need for neuromuscular blockade and sedation, improved venous return and a better ventilation/perfusion (V/Q) matching. For this reason, APRV has been considered a tempting mode of ventilation during acute respiratory failure within the concept of open lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill trauma patients need mechanical ventilation

Exclusion Criteria:

* Pregnant patient.
* Air leak from the chest tube.
* Patient with body temperature > 39 Celsius.
* Acute hepatitis or severe liver disease (Child-Pugh class C).
* Left ventricular ejection fraction less than 30%.
* Heart rate less than 50 beats/min.
* Second or third-degree heart block.
* Systolic pressure < 90 mmHg despite of infusion of 2 vasopressors.
* Patients with known endocrine dysfunction.
* Patient with hypothermia
* Patient on Positive end expiratory pressure more than 14 cmH2o

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
energy expenditure | 48 hours after enrollment
  energy expenditure will be measured using indirect calorimetry via a metabolic module on General Electric ventilator

SECONDARY OUTCOMES:
arterial oxygen tension | 48 hours after enrollment
  measured from arterial sample
arterial carbon dioxide tension | 48 hours after enrollment
  measured from arterial sample
arterial pH | 48 hours after enrollment
  measured from arterial sample

IPD SHARING:
Plan to Share IPD: No